CLINICAL TRIAL: NCT03724630
Title: The Results of Multiple Aspirations and Injections of Unicameral Bone Cyst by Methyl Prednisolone Acetate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, michael moured, principal investigator, Assiut University
Other Study IDs: Assuit University 8000
Record Dates: First submitted 2018-05-15; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-05

CONDITIONS: Simple Bone Cyst
MeSH Terms: conditions — Bone Cysts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the efficacy of methyl prednisolone injection in treatment o f simple bone cyst to prevent all possible complications as pathological fractures and to avoid prolonged restriction of physical activity

DETAILED DESCRIPTION:
unicameral bone cysts (UBCs) are benign, fluid-filled cavities that develop in tubular and flat bones (eg,humerus, femur). These cysts tend to expand and weaken the local bone,but they are not true neoplasms. In 1876, Virchow1 first described these lesions as cystic structures caused by abnormalities in local circulation.

UBCs are also known as simple or solitary bone cysts. They occur almost exclusively in children and adolescents (up to 85% of cases), with a reported peak between ages 3 and14 years and the average age at diagnosis being 9 years.

These lesions represent approximately 3% of all bone tumors and occur more commonly in boys than in girls (2:1). Several treatment options exist for unicameral bone cysts (UBCs), including observation, steroid injection, bone marrow injection, and Surgical procedures have ranged from simple curettage with autologous bone graft or allograft to sub periosteal resection with internal fixation and grafting

.Treatment by multiple injection of steroids produce minimal surgical approach, no hospital stay, and very low morbidity. Three or four injections over a period of 12 month may be enough

ELIGIBILITY:
Inclusion Criteria:

* age .: all children eighteen years of age or younger with unicameral bone cyst
* Patient with previous fracture on top of unicameral bone cyst

Exclusion Criteria:

* patient age more than 18 years old
* patients with malignant tumors
* patients on chronic steroid treatment
* pregnancy

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Each patient will receive a maximum of three or four injections, with at least three months between injections. The indication for a second or third injection will be based on the surgeon's judgment regarding whether the cyst will be healed or not..
  Injections will be performed with the patient under general anesthesia. Under image intensifier. The diagnosis of a unicameral bone cyst will be confirmed by needle aspiration of clear or straw-colored fluid.
  * Methylprednisolone acetate, 3 mg/cm3 of cyst volume with amaximum dose of 180 mg will be injected into the cyst .
  If the cyst was multilocular, each cavity will be injected separately follow up of patients by radiological and clinical outcomes
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
radiological healing of simple bone cyst | one month after injection
  1. Modified Neer classification
     1. Healed cyst : Cyst filled by new bone, with or without small radiolucent area(s) < 1 cm in size
     2. Healing with defect: Radiolucent area(s) < 50% of the diameter of bone, with enough cortical thickness to prevent fracture
     3. Persistent cyst: Radiolucent area > 50% of diameter of the bone and with a thin cortical rim. No increase in the size of the cyst. Continued restriction of activity or repeated treatment is required
     4. Recurrent cyst: Cyst reappeared in a previously obliterated area, or a residual radiolucent area has increased in size
  2. the cyst index which predict the risk of pathological fracture .The cyst index can be calculated as the area of the cyst divided by the square of the diaphysis diameter cyst index equal to or greater than 3.5 indicates a high fracture risk

SECONDARY OUTCOMES:
improvement of symptoms | one month after injection
  clinical healing by asking the patient or his relevant about improvement of symptoms

IPD SHARING:
Plan to Share IPD: Undecided
radiological follow up of patients after one month of injection follow up again by x.ray after three months clinical outcome of patients after injection by visual analogue scale of pain

REFERENCES:
- [Background] Al-Aubaidi Z, Pedersen NW. A bone cyst treated with corticosteroid installation in an osteopetrotic child. J Pediatr Orthop. 2010 Mar;30(2):206-7. doi: 10.1097/BPO.0b013e3181cfcd63. PMID 20179571
- [Background] Pavone V, Caff G, Di Silvestri C, Avondo S, Sessa G. Steroid injections in the treatment of humeral unicameral bone cysts: long-term follow-up and review of the literature. Eur J Orthop Surg Traumatol. 2014 May;24(4):497-503. doi: 10.1007/s00590-013-1211-4. Epub 2013 Apr 3. PMID 23549913
- [Background] Canavese F, Wright JG, Cole WG, Hopyan S. Unicameral bone cysts: comparison of percutaneous curettage, steroid, and autologous bone marrow injections. J Pediatr Orthop. 2011 Jan-Feb;31(1):50-5. doi: 10.1097/BPO.0b013e3181ff7510. PMID 21150732
- [Background] Wright JG, Yandow S, Donaldson S, Marley L; Simple Bone Cyst Trial Group. A randomized clinical trial comparing intralesional bone marrow and steroid injections for simple bone cysts. J Bone Joint Surg Am. 2008 Apr;90(4):722-30. doi: 10.2106/JBJS.G.00620. PMID 18381307
- [Background] Yilmaz G, Aksoy MC, Alanay A, Yazici M, Alpaslan AM. [Treatment of simple bone cysts with methylprednisolone acetate in children]. Acta Orthop Traumatol Turc. 2005;39(5):411-5. Turkish. PMID 16531698
- [Background] Goel AR, Kriger J, Bronfman R, Lauf E. Unicameral bone cysts: treatment with methylprednisone acetate injections. J Foot Ankle Surg. 1994 Jan-Feb;33(1):6-15. PMID 8161995
- [Background] Rud B, Pedersen NW, Thomsen PB. Simple bone cysts in children treated with methylprednisolone acetate. Orthopedics. 1991 Feb;14(2):185-7. doi: 10.3928/0147-7447-19910201-15. PMID 2008387
- [Background] Farber JM, Stanton RP. Treatment options in unicameral bone cysts. Orthopedics. 1990 Jan;13(1):25-32. doi: 10.3928/0147-7447-19900101-06. PMID 2300515